CLINICAL TRIAL: NCT06929676
Title: Assessment of Tooth Mobility After Non-surgical Periodontal Treatment Followed by Tooth Splinting
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Full Professor, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86301125.4.0000.5418
Record Dates: First submitted 2025-03-31; First posted 2025-04-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: periodontal diseases; Tooth Mobility; Periodontal Splints
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Tooth Mobility | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth Mobility Assessment (Experimental): Evaluation of dental mobility before and after non-surgical periodontal treatment, after stabilization by periodontal splints.
  Interventions: Procedure: Periodontal Treatment; Other: assessment of tooth mobility before and after periodontal treatment; Other: Evaluation of Clinical Parameters

INTERVENTIONS:
Procedure: Periodontal Treatment — Non-surgical periodontal treatment with scaling and root planing and dental splinting
Other: assessment of tooth mobility before and after periodontal treatment — Evaluation of dental mobility with a customized device before and after non-surgical periodontal therapy and after stabilization by periodontal splints
Other: Evaluation of Clinical Parameters — Periodontal: probing depth, bone loss, CAL (clinical attachment level) Clinical: occlusal prematurities and collection of gingival crevicular fluid Questionnaire: quality of life (OHIP-14)

SUMMARY:
This clinical study aims to investigate changes in tooth mobility after non-surgical periodontal treatment in anterior teeth with mobility. Twenty patients from the Piracicaba Dental School - Unicamp, diagnosed with stage III or IV periodontitis and grade 2 or 3 tooth mobility, will be selected. Mobility will be assessed using an innovative method involving a customized plate and a tensiometer adapted to apply controlled force.

Initially, participants will undergo a detailed clinical examination, including periodontal evaluation, occlusal analysis, and gingival crevicular fluid collection. After periodontal treatment, which will involve scaling and root planing, mobility will be reassessed after 60 days. Then, a temporary fiber-reinforced resin splint will be applied to the affected teeth and maintained for another 60 days. At the end of the period, the splint will be removed, and new assessments will be conducted.

The study will also analyze the impact of treatment on patients' quality of life (OHIP-14) and the levels of bone and inflammatory markers (OPG, RANK/RANKL, IL-1β, and TNF-α). The findings are expected to provide a better understanding of the response of mobile teeth to periodontal treatment and the role of splinting in stabilizing periodontal tissues.

DETAILED DESCRIPTION:
Study Location and Participants

The study will be conducted at the Specialization Clinic of the Piracicaba Dental School (FOP-Unicamp). Participants will be voluntary patients receiving clinical care at the Undergraduate Clinic of FOP, diagnosed with stage III or IV periodontitis with grades A, B, or C (Papapanou et al., 2018). The inclusion criteria are: periodontal pockets ≥ 4 mm, anterior teeth with mobility (grade 2 or 3) and periodontal attachment loss, and participants of both sexes aged 18 years or older.

All participants will receive treatment in the sextant of the affected tooth/teeth by the researcher, while periodontal treatment of the remaining sextants will be performed as part of the activities of the Undergraduate Clinic at FOP.

Procedure Phase 1: Assessment of Mobility, Clinical Parameters, and Bone Markers Before Non-Surgical Periodontal Treatment Clinical Parameters Initially, volunteers will receive information regarding the etiology and pathogenesis of periodontal diseases. A detailed periodontal evaluation will be performed on the affected sextant (2/5), assessing probing depth (PD) and clinical attachment level (CAL) at six sites per tooth using a calibrated periodontal probe (PCP-UNC 15 tip, Hu-Friedy, Chicago, IL). A complementary periapical radiographic examination will be performed (regions 13-23/33-43), along with the administration of the OHIP-14 questionnaire.

Fabrication of the Tooth Mobility Assessment Device Customized Tray Plate A customized tray plate will be fabricated using Polyethylene Terephthalate Glycol (PET-G) (Bio-Art; Bio-Art Soluções Inteligentes), based on a plaster model of the patient's dentition with a thickness of 1.0 mm. A 3 mm resin layer will be applied over the mobile tooth in the plaster model, creating space on the buccal, lingual/palatal, and incisal surfaces. Relief areas will be made in the acetate plate on the surfaces of mobile teeth, in a circular shape, with diameters larger than 10 mm to allow for displacement force application and measurement.

Instrumentation - Displacement Measurement The instrument chosen and adapted for this research is the Orthodontic Tensiometer (Morelli Orthodontics, Sorocaba/SP, Brazil). Force measurements are presented in gram-force (gf), ranging from 25 gf to 250 gf, with additional readings of 6.25 gf and 12.5 gf. The adapted instrument has a calibration certificate with a precision margin of ±10%, as in the original model.

Displacement will be measured in millimeters using the Absolute digital caliper (Mitutoyo, Illinois, USA), an instrument with a resolution of 0.01 mm/0.0005" and accuracy of ±0.03 mm/0.0015". Measurements will be marked using a silicone stop attached to the millimeter probe, where the instrument tip will touch the dental surface, and the stop will be moved to the external part of the plate on the buccal and lingual/palatal surfaces.

The use of the tensiometer in this study allows for the application of a specific and constant force for each tooth, which will be determined during the initial assessment.

Evaluation of Mobility and Clinical Parameters The examiner will assess the periodontal data of mobile teeth using the PCP-UNC 15 probe (Hu-Friedy), measuring PD and CAL at six sites per tooth. Premature contacts and occlusal interferences will be evaluated using articulating paper. The OHIP-14 questionnaire will be administered, followed by the adaptation of the acetate plate to the patient's arch to assess tooth mobility.

The examiner will apply buccal-lingual and buccal-palatal displacement forces using the tensiometer, determining the force necessary to achieve displacement. A minimum 1-minute interval will be observed between measurements to allow for periodontal ligament relaxation (Konermann et al., 2017). This relaxation time was selected based on investigations into stress relaxation during tooth loading (Komatsu, 2010).

Three measurements will be taken: initial, anterior deflection, and posterior deflection. The initial measurement will be subtracted from the displacement values. All measurements will be performed by the same examiner. Mobility will then be classified according to Lindhe and Nyman (1975), summing the anterior and posterior deflection values.

The displacement force value for each tooth will be specific to each patient and will serve as a standard for mobility reassessments throughout the study.

Gingival Crevicular Fluid Collection Gingival crevicular fluid (GCF) will be collected from each site using sterile absorbent paper cones, which will be carefully inserted into the gingival sulcus at the selected sites. The cone will remain in position for 30 seconds before samples are stored at -20°C in sterilized tubes.

Phase 2: Non-Surgical Periodontal Therapy This phase will involve non-surgical periodontal treatment, including patient visits for mechanical debridement sessions.

Plaque-retentive factors will be eliminated. Supragingival scaling (RDS) of the affected sextant will be performed using Gracey curettes and an ultrasonic scaler (Cavitron® Select) with tips for supragingival use.

Oral hygiene instructions (OHI) will be provided. Supragingival scaling will be performed as needed throughout the study, with careful handling of mobile teeth.

After 15 days, subgingival scaling and root planing (RD/AR) will be performed on sites with periodontal pockets.

Instrumentation will be carried out using Gracey curettes, Mini-Five Gracey curettes, and the Cavitron® Select ultrasonic scaler with tips for both supragingival and subgingival instrumentation. If necessary, occlusal adjustments will be performed on mobile teeth.

Oral hygiene instructions (OHI) will be reinforced at each follow-up visit, which will occur monthly until the study's conclusion.

Phase 3: Reassessment of Tooth Mobility and Clinical Parameters Sixty days after the non-surgical periodontal treatment, tooth mobility will be reassessed using the previously fabricated customized instrument. The same displacement force applied during the initial evaluation will be used for each specific tooth.

If displacement occurs, it will be measured in millimeters and converted into mobility grades according to Lindhe and Nyman (1975), summing the anterior and posterior deflection values.

Clinical parameters will be reassessed, including PD and CAL, which will be measured at six sites per tooth using the PCP-UNC 15 probe (Hu-Friedy). The OHIP-14 questionnaire will be re-administered. GCF samples will be collected again, following the same protocol, and stored at -20°C in sterilized tubes.

Phase 4: Splinting After non-surgical periodontal therapy, all patients will receive a fiber-reinforced composite resin splint (Interlig®, Angelus, 2016), following the manufacturer's instructions.

Clinical Procedure:

Isolation: Absolute isolation of the test tooth and adjacent teeth. Wedge Placement: Interproximal wedges. Surface Preparation: 37% phosphoric acid etching for 30 seconds, adhesive application, light-curing for 20 seconds per segment.

Resin Layer: First composite resin layer applied to lingual/palatal surfaces, followed by adaptation of Interlig fiber and light-curing for 20 seconds per segment.

Final Resin Layer: Applied to cover the fiber, light-cured for 20 seconds per segment.

Finishing and Polishing: Fine diamond burs to remove excess resin and polishing with sequential-grit finishing discs.

Occlusal Adjustment: If premature contacts are present. The splint will remain in place for 60 days, after which all clinical parameters will be reassessed, including radiographic examination.

Analysis of Bone Markers

GCF samples will be collected at three time points:

Baseline 60 days after non-surgical treatment 60 days after splinting removal Bone marker levels (OPG and RANK/RANKL) will be determined using specific kits and MAGpix® technology (MiraiBio, Alameda, CA, USA). These measurements will be analyzed individually using specialized software, with biomarker concentrations expressed in picograms per millimeter (pg/mm)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Stage III and IV Periodontitis (grades A, B and C).
* With periodontal pockets ≥ 4 mm.
* Anterior teeth (13-23 and 33-43) with dental mobility (grade 2 or 3).
* ≥ 18 years old.

Exclusion Criteria:

* Crossbite or edge-to-edge
* Absence of posterior occlusal contact
* Bruxism
* Implants adjacent to the tooth with mobility
* Extreme mobility
* Patients requiring prophylactic antibiotics
* Smokers
* Diabetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of dental mobility with a customized device before and after non-surgical periodontal therapy and after stabilization by periodontal splints | Baseline (Day 0), post- treatment non-surgical periodontal(Day 60), and post splinting (Day 120)
  Tooth mobility will be measured using a custom-made device specifically designed for each patient, allowing for standardized and reproducible assessment. Evaluations will occur at three time points: before the initiation of non-surgical periodontal therapy (baseline), at 60 days (after non-surgical treatment), and at 120 days (after splinting). This method ensures consistent positioning and pressure application during assessments. Each participant will serve as their own control, and the individual tooth will be considered the statistical unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil